CLINICAL TRIAL: NCT02979379
Title: Does Pulmonary Rehabilitation Aggravate or Relieve Symptoms of Pain in Individuals With COPD
Brief Title: Pain in Individuals With COPD During Pulmonary Rehabilitation
Status: Completed | Type: Observational
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, MD, West Park Healthcare Centre
Other Study IDs: 16-001-WP
Record Dates: First submitted 2016-09-01; First posted 2016-12-01 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Pain: Individuals with COPD who experience chronic pain (episodes of daily pain for a duration greater than three months)
  Interventions: Other: Pain
- No Pain: Individuals with COPD who do not experience pain on a regular basis.
  Interventions: Other: Pain

INTERVENTIONS:
Other: Pain

SUMMARY:
This study is aimed at determining the role of pain in individuals with chronic obstructive pulmonary disease (COPD) who are enrolled in a pulmonary rehabilitation (PR) program. It is not known whether pain interferes with an individuals performance in PR, or whether PR aggravates or relieves pain. Individuals with COPD who report chronic pain and those without pain will be enrolled in the study.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a systemic disease associated with dyspnea, fatigue, and poor health-related quality of life. COPD is further complicated by the presence of pain which may be attributed to common comorbidities such as musculoskeletal conditions (osteoarthritis, osteoporosis), cardiac disease or diabetes. Pulmonary rehabilitation (PR) is the cornerstone of treatment for COPD however the impact of pain on PR has not been explored. It is unclear whether those experiencing chronic pain achieve a similar, lesser or greater degree of benefit compared to those without pain, or whether exercise training exacerbates symptoms. Gaining a greater understanding of the effects of an outpatient PR program on pain will provide direction into future specific treatment options which may necessary for managing chronic pain as part of PR.

Individuals with COPD who are beginning an out-patient PR program will be enrolled in the study. Those who report the presence of chronic pain will be classed as the pain group; those who report the absence of chronic pain will be classed as the comparator group. All participants will complete a 6-minute walk test and a Chronic Respiratory Disease Questionnaire (CRDQ) at the beginning of the PR program. These measures will be repeated at the end of the 8-week PR program for all participants. All participants will be asked to report their level of pain using a visual analogue scale every two weeks during the PR program.

Participants reporting chronic pain will also complete a series of questionnaires regarding their pain and coping strategies. These include; the Brief Pain Inventory (BPI), Coping Strategies Questionnaire (CSQ), Fear Avoidance Behavior Questionnaire (FABQ), Hospital Anxiety and Depression Scale (HADS) and Centre for Epidemiological Studies for Depression Survey (CES-D).

ELIGIBILITY:
Inclusion Criteria:

* individuals with moderate to severe COPD based on international (GOLD) criteria
* clinically stable
* no history of acute exacerbation in the past 6 weeks
* able to provide their own informed consent
* referred to out-patient pulmonary rehabilitation at West Park Healthcare Centre

Exclusion Criteria:

* primary diagnosis other than COPD
* known cognitive impairment that would interfere with completing surveys
* cardiac, neurological or orthopedic conditions which prevent the ability to undertake exercise safely

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with moderate to severe COPD enrolled in an out-patient pulmonary rehabilitation program
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Change in qualities of pain (intensity, location, interference) | Change from Baseline to end of 8-Week PR program

SECONDARY OUTCOMES:
Change in coping ability specific to pain and fear avoidance | Change from Baseline to end of 8-Week PR program
Relationship between depression and other psychological factors influencing chronic pain, including coping ability and fear avoidance behaviour | Change from Baseline to end of 8-Week PR program
Change in functional exercise capacity and health related quality of life between those with chronic pain and those without pain | Change from Baseline to end of 8-Week PR program

CONTACTS AND LOCATIONS:
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada